CLINICAL TRIAL: NCT06079502
Title: Electrical Muscle Stimulation Versus Resistive Training On Physical Measures, And Fatigue In Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Ibrahim Yacoub, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Asmaa_Yacoub
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hemodialysis; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation group (Experimental): Thirty patients will receive a supervised program of intradialytic NMES two times per week for 16weeks with medical treatment.
  Interventions: Device: Neuromuscular Electrical Stimulation
- resistive training group (Experimental): Thirty patients will receive a supervised program of intradialytic resistive training two times per week for 16weeks with medical treatment.
  Interventions: Other: resistive training program

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — A supervised program of intradialytic NMES of the quadriceps and calf muscles of both lower limbs with different phases, types and current intensity. The electrical stimulation program will included (total time, intensity, contraction-relaxation phase time): a toning program in the first two weeks.
  Arms: Neuromuscular Electrical Stimulation group
Other: resistive training program — Part one: Warming up for 5 minutes in the form of lower limbs range of motion (active free) exercise from supine position.
  Part two: The main part is the resistive training for quadriceps and calf muscles from supine position using weights in the form of sand bags for 20 min.
  Part three: Cooling down for 5 minutes in the form of lower limbs range of motion (active free) exercise from supine position.
  The training parameters:
  The exercise training will be done during the first 2 hours of HD session using free leg weights. The patient will assume a supine lying position on the treatment plinth and perform the exercises for every lower limb separately while the other limb will be supported on the plinth by therapist or the patient himself. Resistance will be placed at the malleoli level in the distal third of the leg.
  Arms: resistive training group

SUMMARY:
The aim of this study is to compare effect of intradialytic NMES versus resistive training on physical measures and fatigue in HDP.

DETAILED DESCRIPTION:
In this study we will compare between the effect of intradialytic neuromuscular electrical stimulation and resistive training on physical measures, dialysis efficiency and fatigue in HDP. This is first study that will compare between NMES and resistive training in HDP, investigating their effect on physical performance; dialysis efficiency and level of fatigue as previous studies show effect of each intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, with CKF on HD for more than 3 years.
* Age between 40 to 55 years old.
* BMI is between 25 and 29.9 kg/m2.

Exclusion Criteria:

Patients who have one of the following contraindications to the interventions or affect the results

* Cognitive impairment that prevented them from performing the evaluations and who were unable to understand and sign the written informed consent.
* Stroke
* Smokers
* Anemic patients
* Osteoarticular or disabling musculoskeletal disorders
* Uncontrolled hypertension (systolic blood pressure>230 mm Hg and diastolic blood pressure>120 mm Hg)
* Patients with coronary artery disease or heart failure.
* Diabetic patients
* Infectious diseases and chest diseases
* Active smokers' patients with peripheral vascular disease in the lower limbs such as deep vein thrombosis or thromboangiitis

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in maximal strength of quadriceps and calf muscles | at baseline and after 16 weeks of intervention
  By using a Hand held dynamometer: A Kern-type standardized traction dynamometer (Kern CH50 50KG dynamometer) will used to assess the maximal strength of quadriceps and calf muscles will estimate. The patient will remain seated in a fixed chair so the back will supported on the back rest with the hip and knee at 90°, the subject will be asked to exert the greatest possible force without holding the chair with his/her arms,the values of muscular strength variables will be the mean of 3 consecutive measurements obtained by the same investigator to minimize errors
Assessing the change in predicted peak vo2 max | at baseline and after 16 weeks of intervention
  By using a 6-minute walk test (6MWT): It consisted of measuring the maximum distance covered during a 6 min period at an active pace, along a 20 m corridor near the HD unit. At the end of the test period, the total distance travelled was recorded by means of a standardized odometer,that will be used to calculate predicted peak vo2 by using the following equation Mean Peak VO2( ml /kg/min)= 4. 948+ 0. 023*Mean 6 MWD (meters) (SEE 1.1 ml/ kg/ min), standard error of estimate (SEE).

SECONDARY OUTCOMES:
Assessing the change in physical and psychological fatigue | at baseline and after 16 weeks of intervention
  Chalder Fatigue Questionnaire (CFQ11): is a short questionnaire, phrased in simple English with a straightforward answering system, it provides a brief tool to measure both physical and psychological fatigue. It consists from 11 items are answered on a 4-point scale ranging from the asymptomatic to maximum symptomology, a score of 0, increasing to 1, 2 or 3 as they become more symptomatic. The respondent's global score can range from 0 to 33. The global score also spans two dimensions physical fatigue (measured by items 1-7) and psychological fatigue (measured by items 8-11)
Assessing the change in Dialysis efficiency | at baseline and after 16 weeks of intervention
  At baseline and 16 weeks after the intervention, blood samples will be collected after at least 12 h of fasting, and before the HD session, from an antecubital vein via venipuncture. Dialysis efficiency (represented using Kt/V) will be calculated from body weight and blood urea nitrogen (BUN) levels before and after dialysis using the Daugirdas formula as follows. Single-pool Kt/V will be calculated monthly using urea kinetic modeling equations derived from the following equation: (post: pre-dialysis plasma BUN ratio to estimate k. T/v and npcr: mathematical modeling) (second-generation logarithmic estimates of single-pool variable volume kt/v: an analysis of error). Kt/V = - ln(R - 0.008 × t) + [(4-3.5 × R) × UF/W], where R is the ratio of post-dialysis to pre-dialysis serum BUN concentration, t is the duration of hemodialysis in hours, UF is the amount of ultrafiltration (in l) during the HD session, and W is the post-dialysis weight (in kg).

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Yacoub, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided